# Online Study of the Effects of Sugary Drink Warning Labels on Consumption

NCT05079477

2021-08-24

**IRB Study Protocol and Analysis Plan** 

# **Protocol**

# **Objectives**

# Overall objectives

The study objective is to determine to what degree sugar-sweetened beverages (SSB) warning labels increase consumers knowledge about the potential health harms of SSBs and reduce SSB intake. The study aims to assess the impact on purchasing behavior among adults of repeated exposure to SSB warning labels over time.

#### **Background**

Sugar-sweetened beverages (SSBs) significantly contribute to adult and childhood obesity: Nationally, two-thirds of adults and one-third of children are overweight or obese, with higher prevalence among Hispanics and blacks relative to whites (1,2). Excess weight is associated with numerous negative health, psychological, and economic consequences (3-9). No one food or beverage is solely responsible for obesity, but there are several reasons to target SSBs with policy interventions. Sugar-sweetened beverages are drinks with added caloric sweetener (e.g., soft drinks, fruit drinks, sports drinks, and flavored waters containing added sugars), and their consumption is strongly associated with obesity and obesity-related health problems, such as type 2 diabetes and cardiovascular disease (10-18). Intake of SSBs has increased dramatically in the last several decades, and they now represent the largest source of added sugar in the American diet (19,20,42). SSBs are consumed at least once per day by 51% of adults and 64% of youth (43). Although soda consumption has recently declined modestly (44), consumption of other SSBs like sports drinks has increased (19), and todays overall level of SSB consumption remains disturbingly high (19,43). Further, Black and Hispanic individuals consume more kilocalories (kcals) from SSBs compared to white individuals (19). For these reasons, it is important to study interventions to reduce SSB intake among racially and ethnically diverse adults and children.

Nutrition labeling widely used by policy makers, but label design affects degree of impact: Mandatory and voluntary front-of-pack or shelf-tag nutrition labeling systems have been implemented in over 20 countries (45). In the U.S., calories per bottle labels now appear on the front of most beverages (46) and chain restaurants soon must display kcal information on menus (47). Recently, legislative bills were introduced in California (21), New York State (22), Baltimore (23), and San Francisco (24) to require SSBs to display health warning labels on product containers and/or advertisements, much like tobacco warning labels. These warning labels are meant to educate consumers about the potential health harms of over-consuming SSBs and reduce consumption. A number of studies have shown that well-designed nutrition labels can influence behavior (48-58). Examples include: posters displaying SSB calories as minutes required to burn off the calories were associated with reductions in SSB corner store purchases among low-income adolescents (49). Traffic light labels have been associated with sustained decreases in unhealthy item sales and increases in healthy item sales in a hospital cafeteria (50). A randomized-controlled trial found that both traffic light and calorie labels encouraged 10% fewer calories purchased when employees ordered lunch ahead of time through an online portal (51). Supermarket studies have also found that front-of-package and shelf-tag labels influenced purchasing habits (52-58). Overall, food labels can influence behavior, but the design of the label matters.

Effects of tobacco warning labels on knowledge and behavior: The evidence to date suggests tobacco graphic warnings can impact smoking behavior (28-33). Studies across four countries observed significant increases in calls to national telephone helplines after contact information was displayed within health warnings (28-33) and Canada saw a 6% drop in adult smoking prevalence following implementation of graphic warning labels (but graphic labels were introduced along with other tobacco control measures, making it difficult to isolate the independent effect of labels) (34). Research also shows that labels influence beliefs and intentions (25,27,59-65). Smokers in Australia were more likely to think about quitting and avoiding cigarettes after the implementation of large pictorial warnings (59). Significant proportions of smokers surveyed in countries with health warning labels have reported that the labels have motivated them to quit and/or influenced their behavior (60-66). One-fifth of Canadian (65) and twothirds of Australian (62) non-smoking youth reported that warnings helped prevent them from starting to smoke and approximately 90% of U.K. non-smoking youth reported that the warnings deterred them from smoking (61). Mechanisms of label influence: Research shows that tobacco graphic warning labels are more impactful than text labels (59,64,67-78) and both are more impactful than no label (25-33). Pictorial warnings are more effective than text warnings at increasing message salience, awareness, perception of smoking risks, and smokers desire to quit as well as preventing non-smokers from imitating (59,64,66-78). Graphic labels may be more effective than text because they elicit greater emotional reactions. Negative emotional reactions have been associated with increases in thinking about risks, intentions to quit, and quitting behaviors (66,70,75,79). Research also found that warnings depicting shocking images (e.g., rotten teeth, throat, mouth, or lung cancer, gangrenous foot, sick baby in a hospital) were rated as most effective and were more likely to be recalled by smokers (29,66,72,74-76,78,80-83). In addition, accompanying factual information written in a clear and direct manner increases message acceptance (66,72,76,84). While graphic labels with shocking images may be more effective than text-only labels, we decided to test sugar graphic warning labels which factually depict how much sugar is in each beverage. We are testing factual sugar graphic warning labels because they are more legally feasible than shocking images, capture attention, are easy to understand, and inform participants about the potential health risks of consuming added sugars. For these reasons, we hypothesize that sugar graphic warning labels will be more impactful than the caloric control condition. Significant contributions of the proposed research: We expect this research to provide the first causal data on the influence of SSB warning labels relative to standard kcal labels on purchasing and consumption behaviors. These data are much needed as warning label policies have been proposed in two U.S. states and two cities with little empirical evidence. The proposed work will provide an evidence base on the effects of such labels to guide both scientific inquiry and policymaking.

- 1. Flegal KM, Carroll MD, Kit BK, Ogden CL. Prevalence of obesity and trends in the distribution of body mass index among US adults, 1999-2010. JAMA 2012;307:491-7.
- 2. Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity and trends in body mass index among US children and adolescents, 1999-2010. JAMA 2012;307: 483-90.
- 3. Pi-Sunyer FX. The obesity epidemic: pathphysiology and consequences of obesity. Obes Res 2002; 10(Suppl 2): 97S-104S.
- 4. Freedman DS, Khan LK, Dietz WH, Srinivasan SR, Berenson GS. Relationship of childhood obesity to coronary heart disease risk factors in adulthood: the Bogalusa Heart Study. Pediatrics 2001;108(3):712-8.
- 5. Wang CY, McPherson K, Marsh T, Gortmaker SL, Brown M. Health and economic burden of the projected obesity trends in the USA and the UK. The Lancet 2011; 378: 815-25.
- 6. Dietz WH. Childhood weight affects adult morbidity and mortality. J Nutr 1998;128(2 Suppl):411S-4S.
- 7. Kopelman PG. Obesity as a Medical Problem. Nature 2000;404:635-43.
- 8. Puhl RM, Heuer CA. Obesity stigma: important considerations for public health. Am J Public Health 2010; 100: 1019-28.
- 9. Finkelstein EA, Ruhm CJ, Kosa KM. Economic causes and consequences of obesity. Annu Rev Public Health 2005;26:239257.
- 10. Hu FB. Resolved: there is sufficient scientific evidence that decreasing sugar-sweetened beverage consumption will reduce the prevalence of obesity and obesity-related diseases. Obesity Reviews 2013;14:606-19.
- 11. Malik VS, Willett WC, Hu FB. Sugar-sweetened beverages and BMI in children and adolescents: reanalyses of a meta-analysis. Am J Clin Nutr 2009;89:438-9.
- 12. Dong D, Bilger M, van Dam RM, Finkelstein EA. Consumption of specific foods and beverages and excess weight gain among children and adolescents. Health Aff (Millwood) 2015;34:1940-8.
- 13. Ludwig DS, Peterson KE, Gortmaker SL. Relation between consumption of sugar-sweetened drinks and childhood obesity: a prospective, observational analysis. Lancet 2001;357:505-8.
- 14. Ebbeling CB, Feldman HA, Chomitz VR, Antonelli TA, Gortmaker SL, Osganian SK, Ludwig DS. A randomized trial of sugar-sweetened beverages and adolescent body weight. N Engl J Med 2012;367:1407 16.
- 15. de Ruyter JC, Olthof MR, Seidell JC, Katan MB. A trial of sugar-free or sugar-sweetened beverages and body weight in children. N Engl J Med 2012;367:13971406.
- 16. Marshall TA, Levy SM, Broffitt B, Warren JJ, Eicheberger-Gilmore JM, Burns TL, Stumbo PJ. Denta caries and beverage consumption in young children. Pediatrics 2003;112(3, pt 1):e184-e191.
- 17. Marshall TA, Broffitt B, Eichenberger-Gilmore J, Warren JJ, Cunningham MA, Levy SM. The roles of meal, snack, and daily total food and beverage exposures on caries experience in young children. J Public Health Dent 2005;65:166-73.
- 18. Bowen WH, Lawrence RA. Comparison of the cariogenicity of cola, honey, cow milk, human milk, and sucrose. Pediatrics 2005;116:921-6.
- 19. Han E, Powell LM. Consumption patterns of sugar-sweetened beverages in the United States. J Acad Nutr Diet 2013;113:43-53.
- 20. National Cancer Institute. Sources of calories from added sugars among the US population, 2005-06. Risk Factor Monitoring and Methods Branch Web site. Applied Research Program. Mean intake of added sugars & percentage contribution of various foods among U.S population.
- http://appliedresearch.cancer.gov/diet/foodsources/added sugars/table1a.html. (Accessed Jan 20 2016).
- 21. California Senate Bill-1000. Public Health: sugar-sweetened beverages: safety warnings. Available at: http://leginfo.legislature.ca.gov/faces/billNavClient.xhtml?bill id=201320140SB1000. (Accessed June 2014).

- 22. New York State Assembly Bill 2320-B. Requires sugar-sweetened beverages to be labeled with a safety warning. Available at:
- http://assembly.state.ny.us/leg/?default\_fld=&bn=A02320&term=2015&Summary=Y&Actions=Y&Text=Y&Votes=Y#A02320. (Accessed July 2015).
- 23. Sugar-sweetened beverageswarning labels. City of Baltimore Council Bill 16-0617. Article-Health, Sections 16-101-302: Title 16: Sugar-sweetened beverages.
- https://baltimore.legistar.com/LegislationDetail.aspx?ID=2547410&GUID=BF49C0ED-0647-4625-
- B7AEC2592FCAFD7C&Options=ID%7CText%7C&Search=sugar (Accessed January 2016).180
- 24. Sugar-sweetened beverage warning for advertisements. Ordinance No. 100-15. Article 42, Division 1 Sections 4200-06: Sugar sweetened beverage warning ordinance.
- http://www.sfbos.org/ftp/uploadedfiles/bdsupvrs/ordinances15/o0100-15.pdf
- 25. Fathelrahman AI, Omar M, Awang R, Borland R, Fond GT, Hammond D, Zain Z. Smokers responses towards cigarette pack warning labels in predicting quit intention, stage of change, and self-efficacy. Nicotine Tob Res 2009:11:28-53.
- 26. Borland R, Hill D. Initial impact of the new Australian tobacco health warnings on knowledge and beliefs. Tob Control 1997;6:317-25.
- 27. Hammond D. Health warning messages on tobacco products: a review. Tob Control 2011;20:327-37.
- 28. Cavalcante TM. Labelling and Packaging in Brazil. National Cancer Institute, Health Ministry of Brazil; World Health Organization. http://www.who.int/tobacco/training/success\_stories/en/best\_practices\_brazil\_labelling.pdf (Accessed 12 Apr 2010).
- 29. UK Department of Health. Consultation on the Introduction of Picture Warnings on Tobacco Packs: Report on Consultation, 2007. http://www.dh.gov.uk/en/ Consultations/Responsestoconsultations/DH\_077960 (Accessed 13 Jul 2009).
- 30. UK Department of Health. Consultation on the Introduction of Picture Warnings on Tobacco Pack, 2006. http://www.dh.gov.uk/assetRoot/04/13/54/96/04135496.pdf.
- 31. Willemsen MC, Simons C, Zeeman G. Impact of the new EU health warnings on the Dutch quit line. Tob Control 2002;11:381-2.
- 32. Miller CL, Hill DJ, Quester PG, Hiller JE. Impact on the Australian Quitline of new graphic cigarette pack warnings including the Quitline number. Tob Control 2009;18:235-7.
- 33. Wilson N, Li J, Hoek J, Edwards R, Peace J. Long-term benefit of increasing the prominence of a quitline number on cigarette packaging: 3 years of Quitline call data. N Z Med J 2010;123:109-11.
- 34. Health Canada. Canadian Tobacco Use Monitoring Survey (CTUMS). http://www.hc-sc.gc.ca/hcps/tobac-tabac/research-recherche/stat/ctums-esutc 2008-eng.php (Accessed 13 Jul 2009).
- 35. Bollinger B, Leslie P, Sorensen A. Calorie Posting in Chain Restaurants. Am Econ J Econ Policy 2011;3:91-128.
- 36. Krieger JW, Chan NL, Saelens BE, Ta ML, Solet D, Fleming DW. Menu labeling regulations and calories purchased at chain restaurants. Am J Prev Med 2013;44:595-604.
- 37. Auchincloss AH, Mallya GG, Leonberg BL, Ricchezza A, Glanz K, Schwarz DF. Customer responses to mandatory menu labeling at full-service restaurants. Am J Prev Med 2013;45:710-9.
- 38. Wisdom J, Downs JS, Loewenstein G. Promoting Healthy Choices: Information versus Convenience. Am Econ J Appl Econ 2010;2:164-78.
- 39. Elbel B, Kersh R, Brescoll VL, Dixon LB. Calorie labeling and food choices: a first look at the effects on low-income people in New York City. Health Aff (Millwood) 2009;28:w1110-21.
- 40. Elbel B, Mijanovich T, Dixon LB, Abrams C, Weitzman B, Kersh R, Auchincloss AH, Ogedegbe G. Calorie labeling, fast food purchasing and restaurant visits. Obesity (Silver Spring) 2013;21:2172-9.
- 41. Finkelstein EA, Strombotne KL, Chan NL, Krieger J. Mandatory menu labeling in one fast-food chain in King County. Washington. Am J Prev Med 2011:40:122-7.
- 42. Nielsen SJ, Popkin BM. Changes in beverage intake between 1977 and 2001 (published correction appears in Am J Prev Med 2005;28:413). Am J Prev Med 2004;27:205-10.
- 43. Kit B, Fakhouri T, Park S, Nielsen S, Ogden C. Trends in sugar-sweetened beverage consumption among youth and adults in the United States: 1999 2010. Am J Clin Nutr 2013; 98: 180-8.
- 44. Welsh JA, Sharma AJ, Grellinger L, Vos MG. Consumption of added sugars is decreasing in the United States. Am J Clin Nutr 2011;94:726-34.
- 45. Nutrition labels: Nutrition label standards & regulations on the use of claims and implied claims on foods. 2015. World Cancer Research Fund International. URL: http://www.wcrf.org/int/policy/nourishingframework/nutrition-labels (Accessed July 30, 2015).

- 46. Clear on Calories. American Beverage Association Web site. URL:
- http://www.ameribev.org/nutritionscience/clear-on-calories/ (Accessed July 30, 2015).
- 47. Food labeling; nutrition labeling of standard menu items in restaurants and similar retail food establishments. Final rule. Fed Regist. 2014;79(230):71155-259. Epub 2014/12/17 06:00. PubMed PMID:25507861.
- 48. Seymour JD, Yaroch AL, Serdula M, Blanck H, Khan LK. Impact of nutrition environmental interventions on point-of-purchase behavior in adults: a review. Prev Med 2004;39:S108-36.181
- 49. Bleich SN, Herring BJ, Flagg DD, Gary-Webb TL. Reduction in purchases of sugar-sweetened beverages among low-income Black adolescents after exposure to caloric information. Am J Public Health 2012;102:329-35.
- 50. Thorndike AN, Riis J, Sonnenberg LM, Levy DE. Traffic-light labels and choice architecture: promoting healthy food choices. Am J Prev Med 2014;46:143-9.
- 51. VanEpps EM, Downs JS, Loewenstein G. Calorie Label Formats: Using Numbers or Traffic Lights to Reduce Lunch Calories. Journal of Public Policy & Marketing In-Press.
- 52. Sutherland LA, Kaley LA, Fischer L. Guiding stars: the effect of a nutrition navigation program on consumer purchases at the supermarket. Am J Clin Nutr 2010;91:1090S94S.
- 53. Levy AS, Mathews O, Stephenson M, Tenney JE, Schucker RE The impact of a nutrition information program on food purchases. J Public Policy Mark 1985;4:113.
- 54. Schucker RE, Levy AS, Tenney J, Mathews O. Nutrition shelf-labeling and consumer purchase behavior. J Nutr Educ 1992;24:7581.
- 55. Rodgers AB, Kessler LG, Portnoy B, Potosky AL, Patterson B, Tenney J, Thompson FE, Krebs-Smith SM, Breen N, Mathews O, Eat for Health: a supermarket intervention for nutrition and cancer risk reduction. Am J Public Health 1994;84:726.
- 56. Holmes AS, Estabrooks PA, Davis GC, Serrano EL. Effect of a grocery store intervention on sales of nutritious foods to youth and their families. J Acad Nutr Diet 2012;112:897901.
- 57. Muller TE. The use of nutritive composition data at the point of purchase. J Nutr Educ 1984;16:13741.
- 58. Curhan RC. The effects of merchandising and temporary promotional activities on the sales of fresh fruit and vegetables in supermarkets. J Mark Res 1974;11:28694.
- 59. White V, Webster B, Wakefield M. Do graphic health warning labels have an impact on adolescents smoking related beliefs and behaviours? Addiction 2008;103:1562-71.
- 60. European Commission. Eurobarometer: Survey on Tobacco (Analytical Report). 2009.
- http://ec.europa.eu/public opinion/flash/fl 253 en.pdf (Accessed 12 Apr 2010).
- 61. Moodie C, Mackintosh AM, Hammond D. Adolescents response to text-only tobacco health warnings: Results from the 2008 UK Youth Tobacco Policy Survey. Eur J Public Health 2010;20:463-9.
- 62. Shanahan P, Elliott D. Evaluation of the Effectiveness of the Graphic Health Warnings on Tobacco Product Packaging 2008. Canberra: Australian Government. Department of Health and Ageing,
- 2009.http://www.health.gov.au/internet/main/ publishing.nsf/Content/health-pubhlth-strateg-drugs-tobaccowarnings.htm (Accessed 12 Apr 2010).
- 63. Koval JJ, Aubut JA, Pederson LL, OHegarty M, Chan SS. The potential effectiveness of warning labels on cigarette packages: the perceptions of young adult Canadians. Can J Public Health 2005;96:353-e6.
- 64. Hammond D, Fong GT, Borland R, Cummings KM, McNeill A, Driezen P. Text and Graphic Warnings on Cigarette Packages: Findings from the ITC Four Country Survey. Am J Prev Med 2007;32:202-9.
- 65. Environics Research Group. The Health Effects of Tobacco and Health Warning Messages on Cigarette Packages Survey of Youth: Wave 12 Surveys. Prepared for Health Canada. 2007.
- 66. Hammond D, Fong GT, McDonald PW, Cameron R, Brown KS. Impact of the graphic Canadian warning labels on adult smoking behaviour. Tob Control 2003;12:391-5.
- 67. International Tobacco Control Policy Evaluation Project. FCTC Article 11eTobacco Warning Labels: Evidence and Recommendations from the ITC Project. 2009. http://www.itcproject.org (Accessed 22 Jun 2009).
- 68. Liefeld JP. The Relative Importance of the Size, Content and Pictures on Cigarette Package Warning Messages. Prepared for Health Canada. Guelph, Canada: Department of Consumer Studies, University of Guelph, 1999.
- 69. OHegarty M, Pederson LL, Nelson DE, Mowery P, Gable JM, Wortley P. Reactions of young adult smokers to warning labels on cigarette packages. Am J Prev Med 2006;30:467-73.
- 70. Kees J, Burton S, Andrews JC, Kozup J. Understanding how graphic pictorial warnings work on cigarette packaging. J Public Policy Mark 2010;29:265-76.
- 71. Environics Research Group. Testing New Health Warning Messages for Cigarette packages: A Summary of Three Phases of Focus Group Research: Final Report. Prepared for Health Canada, 2000. http://www.tobaccolabels.ca/healt/canada (Accessed 12 Jul 2009).

- 72. Corporate Research Associates. Creative Concept Testing for Health Warning Messages. Prepared for Health Canada, 2005. http://www.tobaccolabels.ca/healt/ canada2005 (Accessed 13 Jul 2009).
- 73. Clemenger BBDO. Marketing Inputs to Assist the Development of Health Warnings for Tobacco Packaging. Report to the Ministry of Health: Review of the Smoke-free Environments Regulations, 2004.182

http://www.ndp.govt.nz/moh.nsf/indexcm/ndp- publications-marketinginputsmay2006 (Accessed 13 Jul 2009).

- 74. BRC Marketing & Social Research. Smoking Health Warnings Stage 1: The Effectiveness of Different (Pictorial) Health Warnings in Helping People Consider their Smoking-Related Behaviour. Prepared for the New Zealand Ministry of Health, 2004.
- 75. Elliott & Shanahan (E&S) Research. Developmental Research for New Australian Health Warnings on Tobacco Products: Stage 1. Prepared for the Population Health Division Department of Health and Ageing. Commonwealth of Australia. 2002
- http://www.health.gov.au/internet/main/publishing.nsf/Content/474DA5DAC70608F2CA2571A1001C7DFE/\$File/warnings\_stage1.pdf (Accessed 13 Jul 2009).
- 76. Les Etudes de Marche Createc. Final Report: Qualitative Testing of Health Warnings Messages. Prepared for the Tobacco Control Programme Health Canada. 2006.
- 77. Hassan LM, Shiu E, Thrasher JF, Fong GT, Hastings Gerard. Exploring the effectiveness of cigarette warning labels: findings from the United States and United Kingdom arms of the International Tobacco Control (ITC) Four Country Survey. Int J Nonprofit Volunt Sect Mark 2008;13:263-74.
- 78. Wade B, Merrill RM, Lindsay GB. Cigarette pack warning labels in Russia: how graphic should they be? Eur J Public Health 2011;21:366-72.
- 79. Peters E, Romer D, Slovic P, Jamieson KH, Wharfield L, Mertz CK, Carpenter SM. The impact and acceptability of Canadian-style cigarette warning labels among U.S. smokers and nonsmokers. Nicotine Tob Res 2007;9:473-81.
- 80. Devlin E, Anderson S, Hastings G, MacFadyen L. Targeting smokers via tobacco product labellings: opportunities and challenges for Pan European health promotion. Health Promot Int 2005;20:41-9.
- 81. Strahan EJ, White K, Fong GT, Fabrigar L, Zanna M, Cameron R. Enhancing the effectiveness of tobacco package warning labels: a social psychological perspective. Tob Control 2002;11:183-90.
- 82. Gallopel-Morvan K, Gabriel P, Le Gall-Ely M, Rieunier S, Urien Bertrand. The use of visual warnings in social marketing: The case of tobacco. J Bus Res 2011;64:7-11.
- 83. Nascimento BE, Oliveira L, Vieira AS, Joffily M, Gleiser S, Pereira MG, Cavalcante T, Volchan E. Avoidance of smoking: the impact of warning in Brazil. Tob Control 2008;17:405-9.
- 84. Decima Research Testing of Health Warning Messages and Health Information Messages for Tobacco Products Executive Summary. Prepared on behalf of Health Canada, 2009.

### Study Design

#### Design

The primary objective of this study is to determine, before wide-scale implementation, to what degree SSB warning labels increase consumers knowledge about the potential health harms of SSBs and reduce SSB intake. This study will examine how repeated exposure to SSB warning labels influence adults' purchasing behaviors over time. Participants will be blindly randomized to 1 of 2 study conditions. Although participants will not know there are other conditions, it will be impossible to blind them to their own conditions as they will view the labels associated with their conditions.

#### **Study duration**

Participants will be randomized to 1 of 2 conditions and will buy snacks and beverages for four weeks via an online store. We anticipate it will take approximately one year to finish recruiting all subjects and for all subjects to complete the study. We will start recruiting subjects once IRB approval is obtained.

# **Characteristics of the Study Population**

#### Target population

We will recruit 216 racially and ethnically diverse parents from Philadelphia and the surrounding communities. Participants will need to be at least 18 years old, a primary caregiver of a child between the ages of 6 and 11, able to read and speak English, be the primary grocery shopper for their household, have regular Internet access, live in the Philadelphia area (within Amazon Fresh delivery radius), must purchase SSBs at least once per month and report that the oldest of their children between 6 and 11 years old is consuming SSBs at least twelve times per month or

approximately three times a week. Additionally, participants must not have participated in the prior Warning Label Online Store study, or the Beverage Tax Evaluation study conducted by our research team.

# **Subjects enrolled by Penn Researchers**

216

#### **Subjects enrolled by Collaborating Researchers**

n

# **Vulnerable Populations**

Children Form

Pregnant women (if the study procedures may affect the condition of the pregnant woman or

fetus) Form

Fetuses and/or Neonates Form

**Prisoners Form** 

Other

x None of the above populations are included in the research study

The following documents are currently attached to this item:

There are no documents attached for this item.

#### **Subject recruitment**

We will advertise through Craigslist. We will also leverage the resources and community relationships of the UPENN CDC-funded PRC co-directed by Drs. Glanz and Volpp (Co-Is) who both have a long track record of successfully working with local communities on research partnerships. We will also utilize Facebook Advertising through a Facebook page created for the study in order to reach more potential participants throughout the Philadelphia community (Craigslist language and Facebook flyer attached to this submission). Following all guidelines related to the COVID-19 pandemic, we will also hand out flyers directly to consumers and post them in neighborhoods if it is safe to do so.

When individuals call in to inquire about the study, they will be asked a series of questions to determine if they are eligible for the study.

Will the recruitment plan propose to use any Penn media services (communications, marketing, etc.) for outreach via social media avenues (examples include: Facebook, Twitter, blogging, texting, etc.) or does the study team plan to directly use social media to recruit for the research? No

# The following documents are currently attached to this item:

There are no documents attached for this item.

# **Subject compensation\***

Will subjects be financially compensated for their participation? Yes

# The following documents are currently attached to this item:

There are no documents attached for this item.

# If there is subject compensation, provide the schedule for compensation per study visit or session and total amount for entire participation, either as text or separate document

At the start of the study, participants will be given assigned money in the form of a store gift card to which researchers will add money throughout the course of the study. Participants will initially be given \$15 to use to purchase items in the online store. Participants will be asked to purchase at least two items in the store each week (they must select at least one snack and one beverage). After purchasing at least two items during the first week, a participant's account will increase by \$15 the following week as an incentive to remain in the study. For weeks three and four, participants will receive an additional \$17 in their account to purchase more products in the store. Whatever money they do not spend in the online store will accrue over time and at the end of the study, they will be mailed a physical ClinCard (debit card) that will be loaded with the value of the unspent money as well as an additional \$20 for completing the final survey. The total compensation for full participation is \$84 per participant.

# **Study Procedures**

# Suicidal Ideation and Behavior

Does this research qualify as a clinical investigation that will utilize a test article (ie- drug or biological) which may carry a potential for central nervous system (CNS) effect(s)?

No

#### **Procedures**

To conceal the study's purpose, participants will be told that we are conducting consumer market research to learn about their experiencing shopping in an online snack store. Participants will be recruited on the phone. During this initial phone call, consent will be obtained and documented by the research assistant in REDCap, and participants will be given a tutorial about shopping in the online store. After the recruitment call, participants will be texted or emailed a link to a survey asking them to provide demographic information and beverage consumption information in a REDCap survey. They will also be mailed a welcome packet which includes a copy of the informed consent form, a Welcome Letter that gives them an overview of what they will be asked to do as well as answers to any frequently asked questions, in addition to an Online Store Guide to help participants navigate our online store interface (all attached to this submission).

After consent is obtained, participants will be randomized to one of 2 label conditions in REDCap: 1) calorie labels (control); or 2) sugar graphic warning labels. Afterwards, participants will be emailed a web-link and password that will direct them to the store interface based on their label condition. Participants will be asked to shop in the store for a total of four weeks. For the first two weeks, participants will receive \$15 in their online store account. For weeks three and four, participants will receive \$17 in their online store account. For all of the weeks, participants will be asked to purchase at least one beverage and one snack from the online store. Each week participants will receive up to 3 text reminders to shop in the online store. If participants are non-responsive via text, we will send 3 email reminders, and then 3 phone calls. Twice a day (excluding weekends) an RA will process and purchase the orders through our Amazon.com Prime account, which will enable us to ship the actual purchases within a few days. If for some reason Amazon Fresh does not have a product in stock, we will send the participant a replacement item. At the end of four weeks, research assistants will email or text participants with a REDCap link to a final survey for them to complete. After participants complete the final survey, a debriefing and consent form will appear on their screen. After participants read the debriefing statement, they will have the choice of either withdrawing from the study or indicating that it is still okay for the researchers to use their data (see attached). Participants will be required to answer this last question of consent before the survey can be considered completed.

Upon study completion, participants will be mailed a final study packet which includes the following: 1) Study Conclusion Letter (thanks them for their participation and gives a brief overview of the next steps to activate their study debit card in the form of a ClinCard which we will use to pay them for their participation), 2) Study ClinCard and ClinCard FAQ (details information on how to use a ClinCard), 3) Final Debrief Information Sheet (paper copy of the debriefing form that they saw on the Final Survey). All forms are attached to this submission.

# The following documents are currently attached to this item:

There are no documents attached for this item.

#### Deception

Does your project use deception?

Yes

A. Deception/incomplete disclosure is typically only acceptable in studies with no more than minimal risk. Please detail why this study is minimal risk.

This study poses minimal risks. Participants will answer questions over the phone with a research participant, shop in a Shopify store, and complete self-report surveys via REDCap. No protected health information will be collected.

B. The deception/incomplete disclosure should have no adverse effects on welfare. Please outline how all adverse effects are minimized.

One potential risk is breach of confidentiality. We will minimize these risks by assigning a random participant identification number and stripping all identifying information from the dataset at the end of the study. All study data will be stored in REDCap and the PEACH Lab secure drive. Only the researchers involved in this study and those responsible

for research oversight will have access to the identifiable information provided. Any de-identified data shared will be done so via PennBox, a secure method to transfer files.

- C. The IRB must determine that the value of the study is sufficient to warrant waiving some aspects of the requirement for full disclosure in the informed consent process. Please outline the scientific validity for using deception in this instance. There is some information about the study that we will not initially share with participants. It will be necessary to omit certain details on the first day of the study so that we can create a realistic situation that will allow participants to react genuinely and spontaneously without second-guessing their intuitive choices. To conceal the study's purpose, participants will be told that we are conducting consumer market research about online shopping experiences and behaviors. We will explain that the online interface they are using may change throughout the study.
- D. There is no alternative to address the scientific question in a valid manner but to use deception/incomplete disclosure. Other effective, non-deceptive approaches are not feasible. Please detail why alternatives are not feasible. There is some information about the study that we will not initially share with participants. It will be necessary to omit certain details on the first day of the study so that we can create a realistic situation that will allow participants to react genuinely and spontaneously without second-guessing their intuitive choices. To conceal the study's purpose, participants will be told that we are conducting consumer market research about online shopping experiences and behaviors. We will explain that the online interface they are using may change throughout the study.
- E. Debriefing is done, when appropriate, and the deception/incomplete disclosure is explained to the participant before the end of participation in the research. Please detail if you are debriefing participants, and if not, why not. All participants will be debriefed at the end of the study to inform them about the true study purpose. At the end of four weeks, research assistants will text or email participants with a REDCap link to a final survey for them to complete. After participants complete the final survey, a debriefing and consent form will appear on their screen. After participants read the debriefing statement, they will have the choice of either withdrawing from the study or indicating that it is still ok for the researchers to use their data. Participants will be required to answer the last question before the survey can be considered completed.
- F. When appropriate, subjects could be informed prospectively of the use of deception/incomplete disclosure and consent to its use: see the suggested consent language: "In some research studies, the investigators cannot tell you exactly what the study is about before you participate in the study. We will describe the tasks in the study in a general way, but we can't explain the real purpose of the study until after you complete these tasks. When you are done, we will explain why we are doing this study, what we are looking at, and any other information you should know about this study. You will also be able to ask any questions you might have about the study's purpose and the tasks you did. Though we may not be able to explain the real purpose of the study until after you complete the tasks, there are no additional risks to those that have been described in this consent form."

There is some information about the study that we will not initially share with participants. It will be necessary to omit certain details on the first day of the study so that we can create a realistic situation that will allow participants to react genuinely and spontaneously without second-guessing their intuitive choices. To conceal the study's purpose, participants will be told that we are conducting consumer market research about online shopping experiences and behaviors. We will explain that the online interface they are using may change throughout the study.

#### **International Research**

Are you conducting research outside of the United States?

#### **Analysis Plan**

We will use a generalized estimating equation (GEE) modeling approach. Specifically, a linear GEE model of the transformed outcome (log10 (calories +1)) will be fit to a model with 1 categorical variable as the independent variable indicating the experimental condition (e.g., control is the reference) and an indicator for the corresponding measurement time (1, 2, 3, or 4 weeks). Such a model will allow us to examine overall treatment and time effects. Inferences will be adjusted appropriately to control the Type 1 error rate for multiple comparisons (e.g., Bonferroni).